CLINICAL TRIAL: NCT06733142
Title: The Effects of a Commercially Available High Protein Spoonable on Amino Acid Bioavailability in 18-45-year-old Male and Female Volunteers.
Brief Title: Spoonable Bioavailability
Acronym: BOLT_Part A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glyn Howatson (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Sponsor-Investigator, Glyn Howatson, Professor, Northumbria University
Organization: Northumbria University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BOLT_PartA_7911
Record Dates: First submitted 2024-10-25; First posted 2024-12-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-12

CONDITIONS: Amino Acid Absorption; Amino Acid Plasma Profile; Amino Acids, Essential
Keywords: Bioavailability; High Protein; Amino Acids

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Product (Experimental): High protein commercially available spoonable yoghurt (1 serving = 45 g protein comprising 3 yoghurt pots totalling 480 g) (Danone Nutricia).
  Interventions: Dietary Supplement: Test Product: Yoghurt
- Micellar casein drink (Active Comparator): Micellar casein drink (1 serving = 45 g protein/480 g).
  Interventions: Dietary Supplement: Micellar casein drink
- Placebo (Placebo Comparator): Flavoured water-based placebo jelly (1 serving = 0 g protein comprising 3 jelly pots totalling 480 g).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Test Product: Yoghurt — High protein spoonable yoghurt
  Arms: Test Product
Dietary Supplement: Micellar casein drink — Micellar casein drink made from water, casein powder and fruit syrup
  Arms: Micellar casein drink
Dietary Supplement: Placebo — Placebo sugar free jelly
  Arms: Placebo

SUMMARY:
The key research objective is to characterise the amino acid (AA) bioavailability for 4 hours following consumption of a single serving of a high protein spoonable yoghurt, compared to a micellar casein drink or a flavoured water-based placebo jelly, in 18-45-year-old males and females. An additional exploratory objective is to characterise the time to reach peak concentration (Tmax) of AA after consumption of a single serving of each product.

DETAILED DESCRIPTION:
This study is a single-blind, three-way, randomised crossover design. It involves four visits to the laboratory in total; the first session will be a pre-screening and familiarisation, and the subsequent three sessions will be 3 x bioavailability assessments, separated by a washout period of a minimum of 5 days and maximum of 21 days. The bioavailability assessments will be identical except for the product consumed; subjects will receive one serving of the following in a random order:

1. Test product: High protein spoonable yoghurt (1 serving = 45 g protein comprising 3 yoghurt pots totalling 480 g) (Danone Nutricia).
2. Control product 1: Micellar casein drink (1 serving = 45 g protein/480 g).
3. Control product 2: flavoured water-based placebo jelly (1 serving = 0 g protein comprising 3 jelly pots totalling 480 g).

A follow-up communication via telephone will be conducted within 7 days of completion of the fourth and final session to ensure there are no adverse effects of participation.

A detailed overview of the research activity that will take place in each session is provided below:

Visit 1: Pre-screening: Volunteers will receive information on the study, and they will be familiarised with the requirements for participation and provide written informed consent. Subjects will be requested to complete 3-day food and exercise diaries, comprising of 1 weekend day, 1 rest day, and 1 exercise day within a week of the trial. This will be handed in on Visit 2. Subjects' body height, body mass, body composition, and body mass index (BMI) will be measured.

Visits 2-4: Bioavailability assessments: Subjects will refrain from physical activity and alcohol consumption 24 hours before each visit and caffeine 12 hours before each visit. After an overnight fast (at least 10 hours), subjects will come to the lab to participate. Study staff will collect food and exercise diaries from subjects. If the inclusion criteria continue to be met, participants can continue into the trial. A cannula will be inserted into an antecubital vein by a qualified member of the study team, with appropriate standard procedures for cannula care followed throughout the visit duration.

Subjects will consume one serving of one of the study products (~10 minutes). Subjects Blood samples will be drawn at time (T) = 0 min (baseline, before consumption) and at t = 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 min after the study product intake. Throughout the study visits, subjects are not allowed to eat, but will be permitted to drink up to 250 mL of water after the first 2 hours - the volume consumed and timing during Visit 2 will be replicated as best as possible on subsequent visits. In addition, subjects will be asked to abstain from any physical exercise other than incidental walking during the study visits.

Within 5-21 days after Visit 2, volunteers will undergo the same intervention with the second and then third study products at Visits 3 and 4, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 45 years
* Body Mass Index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
* Written informed consent
* Willingness and ability to comply with the protocol in the opinion of the Investigator
* Judged by the Investigator to be in good health as assessed by a health screening questionnaire
* Currently identifies as the same biological sex as at birth

Exclusion Criteria:

* Any known ongoing medical condition that interferes significantly with absorption and digestion and/or gastrointestinal (GI) function (e.g. inflammatory bowel disease, gastroesophageal reflux disease, celiac disease, diaphragmatic hernia or diaphragmatic surgery, gastric ulcer, gastritis, gall bladder problems, pancreatitis, GI cancer, oesophageal and/or gastric surgery), in opinion of the investigator.
* Known musculoskeletal or soft tissue injury
* Known cardiovascular disease, disease related to the immune system and/or the respiratory system
* Known renal or hepatic failure or known thyroid dysfunction
* Known Diabetes Mellitus type I or type II, insulin resistance or metabolic syndrome
* Any ongoing cancer (except for basal cell carcinoma) and/ or cancer treatment
* Known anaemia or low haemoglobin or low iron status
* Any known bleeding disorder or reaction to withdrawal of blood samples
* Use of oral and systemic use of prokinetics, laxatives, antidiarrheals, anticoagulants within 2 weeks prior to screening
* Use of systemic antibiotics within 4 weeks prior to screening
* Any known allergies or intolerances to ingredients of the study product, i.e. cow's milk allergies, lactose intolerance
* Adherence to a strict dietary regime (e.g. vegetarian/ vegan/ paleo/ketogenic/intermittent fasting/ high protein diet (>1.6 g/kg body weight/day) or a weight loss program)
* Use of any nutritional supplements or additional protein supplements or nutritional support within 4 weeks prior to screening
* Falling below or exceeding the classification of Tier 1 or Tier 2 (McKay et al 2022, IJSPP. 17, 317-331). Ranging from minimum of meeting WHO guidelines for physical activity up to training ~3 times per week and local level representation in a sport.
* Known pregnancy and/or lactation
* Current smoking or stopped smoking for <1 month prior to screening (except for incidental smoking of ≤3 cigarettes/cigars/pipes per week on average in the last month)
* Average alcohol use of >21 glasses* per week for men or >14 glasses per week for women (on average during the last 6 months) or drug/ medicine abuse in opinion of the investigator
* Participation in any other clinical study with investigational or marketed products concomitantly or within 4 weeks before screening.
* Major medical or surgical event requiring hospitalization within the preceding 3 months and/or scheduled in the period of study participation relevant in the opinion of the Investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Peak Concentration for Total Amino Acids | At timepoints: T = 0 min (baseline, before consumption) and at t = 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 min after the study product intake.
  Descriptive summary of peak concentration (Cmax) [µM] for total AA after consumption of a single serving of a high protein spoonable yoghurt, micellar casein drink, and flavoured water-based placebo jelly in 18-45-year-old males and females over 4 hours.
Incremental Area Under Curve for Total Amino Acids | At timepoints: T = 0 min (baseline, before consumption) and at t = 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 min after the study product intake.
  Descriptive summary of incremental area under the curve (iAUC) [µM] for total AA after consumption of a single serving of a high protein spoonable yoghurt, micellar casein drink, and flavoured water-based placebo jelly in 18-45-year-old males and females over 4 hours.

SECONDARY OUTCOMES:
Time to Reach Maximum Concentration of Amino Acids | At timepoints: T = 0 min (baseline, before consumption) and at t = 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 min after the study product intake.
  Descriptive summary of time to reach maximum concentration (Tmax) [min] of total AA after consumption of a single serving of a high protein spoonable yoghurt, micellar casein drink, and flavoured water-based placebo jelly in 18-45-year-old males and females over 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513